CLINICAL TRIAL: NCT03110380
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Switching From a Regimen of Dolutegravir and Either Emtricitabine/Tenofovir Alafenamide or Emtricitabine/Tenofovir Disoproxil Fumarate to a Fixed Dose Combination of Bictegravir/ Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected Subjects Who Are Virologically Suppressed
Brief Title: Switching to a Fixed Dose Combination of Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) in Human Immunodeficiency Virus Type 1 (HIV-1) Infected Adults Who Are Virologically Suppressed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-380-4030; 2017-000308-17 (EudraCT Number)
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; emtricitabine tenofovir alafenamide; dolutegravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- B/F/TAF (Experimental): Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) fixed-dose combination (FDC) tablet + dolutegravir (DTG) placebo tablet + emtricitabine/tenofovir alafenamide (F/TAF) placebo tablet administered without regard to food for at least 48 weeks.
  Interventions: Drug: B/F/TAF; Drug: DTG Placebo; Drug: F/TAF Placebo
- DTG + F/TAF (Active Comparator): DTG 50 mg tablet + F/TAF FDC tablet + B/F/TAF placebo tablet administered without regard to food for at least 48 weeks.
  Interventions: Drug: F/TAF; Drug: DTG; Drug: B/F/TAF Placebo
- Open-label Phase B/F/TAF from B/F/TAF (Experimental): Participants who received B/F/TAF in double-blind phase and from a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
  Interventions: Drug: B/F/TAF
- Open-label Phase B/F/TAF from DTG + F/TAF (Experimental): Participants who received DTG + F/TAF in double-blind phase and from a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — 50/200/25 mg FDC tablet(s) administered orally once daily
  Other Names: GS-9883/F/TAF; Biktarvy®
  Arms: B/F/TAF; Open-label Phase B/F/TAF from B/F/TAF; Open-label Phase B/F/TAF from DTG + F/TAF
Drug: F/TAF — 200/25 mg FDC tablet(s) administered orally once daily
  Other Names: Descovy®
  Arms: DTG + F/TAF
Drug: DTG — 50 mg tablet(s) administered orally once daily
  Other Names: Tivicay®
  Arms: DTG + F/TAF
Drug: DTG Placebo — Tablet(s) administered orally once daily
  Arms: B/F/TAF
Drug: F/TAF Placebo — Tablet(s) administered orally once daily
  Arms: B/F/TAF
Drug: B/F/TAF Placebo — Tablet(s) administered orally once daily
  Arms: DTG + F/TAF

SUMMARY:
The primary objective of this study is to evaluate the efficacy of switching from a regimen of either dolutegravir (DTG) and emtricitabine /tenofovir alafenamide (F/TAF) or DTG and emtricitabine/tenofovir disoproxil fumarate (F/TDF) to a fixed dose combination (FDC) of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus DTG+F/TAF in virologically suppressed HIV-1 infected adults with or without antiretroviral (ARV) resistance.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently receiving an ARV regimen of DTG+F/TAF or DTG+F/TDF for the following minimum time periods:

  * ≥ 6 months (if there is documented or suspected nucleoside/nucleotide reverse transcriptase inhibitor (NRTI) resistance prior to the screening visit)
  * ≥ 3 months (if there is no documented or suspected NRTI resistance prior to the screening visit)
* Documented plasma HIV-1 ribonucleic acid (RNA) < 50 copies/mL during treatment with DTG+F/TAF or DTG+F/TDF (for a minimum period of ≥ 6 or ≥ 3 months, as applicable) preceding the screening visit
* Plasma HIV-1 RNA levels < 50 copies/mL at screening visit
* Estimated Glomerular Filtration Rate (eGFR) ≥ 30 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* No documented resistance to integrase stand transfer inhibitors (INSTIs) or confirmed virologic failure
* Eligible adults with chronic hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection are permitted to enroll

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (94):
- United States (66):
  - Spectrum Medical Group, Phoenix, Arizona
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Highland Hospital - Alameda Health System, Oakland, California
  - Cares Community Health, Sacramento, California
  - Kaiser Permanente, Sacramento, California
  - Hepatitis/HIV Clinical Trials Group (HHCTG), San Francisco, California
  - Kaiser Permanente, San Francisco, California
  - Kaiser Permanente, Department of Infectious Diseases, San Leandro, California
  - University of Colorado Denver, University of Colorado Hospital, Aurora, Colorado
  - Whitman-Walker Institute, Washington D.C., District of Columbia
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Providence Hospital Center for Infectious Diseases, Washington D.C., District of Columbia
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary J. Richmond, M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami Divison of Infectious Diseases Clinical Research Unit, Miami, Florida
  - AIDS Healthcare Foundation - South Beach, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AHF-Pensacola, Pensacola, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - St. Joseph's Hospital Comprehensive Research Institute, Tampa, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Emory Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AU Medical Center, Augusta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - John A. Burns School of Medicine, University of Hawaii Clinics at Kaka'ako, Honolulu, Hawaii
  - University of Louisville 550 Clinic, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Community Research Initiative of New England, Boston, Massachusetts
  - Metro West Medical Center, Framingham, Massachusetts
  - Claudia T Martorell, MD., LLC d/b/a The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Abbott Northwestern Hospital part of Allina Health, Minneapolis, Minnesota
  - Hennepin County Medical Center, Positive Care Clinic, Minneapolis, Minnesota
  - Kansas City CARE Clinic, Kansas City, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Prime Healthcare Services - St. Michael's LLC d/b/a Saint Michael's Medical Center, Newark, New Jersey
  - Southwest CARE Center, Albuquerque, New Mexico
  - Southwest CARE Center, Santa Fe, New Mexico
  - North Shore University Hospital/Division of Infectious Diseases, Manhasset, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - NC TraCS Institute - CTRC; University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Heath System, Durham, North Carolina
  - East Carolina University (ECU), The Brody School of Medicine, Adult Specialty Care, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Palmetto Health Richland (Regulatory and Study Supply Shipping), Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - AIDS Arms Inc/ Trinity Health and Wellness Center, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - The Crofoot Research Center, INC (DBA: Gordon E. Crofoot MD PA), Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Peter Shalit, M.D., Seattle, Washington
  - MultiCare Rockwood HIV Critical Care Clinic, Spokane, Washington
- Medizinische Universitat Wien, Universitatsklinik fur Dermatologie, Vienna, Austria
- Canada (6):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Spectrum Health Clinic, Vancouver, British Columbia
  - Winnipeg Regional Health Authority - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Maple Leaf Research / Maple Leaf Medical Clinic, Toronto, Ontario
  - Clinique de Médecine Urbaine du Quartier Latin, Montreal, Quebec
  - Chronical Viral Illness Service/McGill University Health Care (MUHC), Montreal, Quebec
- France (8):
  - Hôpital Saint-André, Bordeaux
  - Hôpital Croix-Rousse, Lyon
  - Hôpital Gui de Chauliac, CHU de Montpellier, Montpellier
  - CHU de Nice-l'Archet, Nice
  - CHU Bichat, Paris
  - AP-HP Hôpital Tenon, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
- Germany (9):
  - zibp Zentrum für Infektiologie Berlin Prenzlauer Berg, Berlin
  - EPIMED Gesellschaft fur epidemiologische und klinische Forschung in der Medizin mbH, Berlin
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I, Klinisches Studienzentrum Immunologie, Bonn
  - Universitätsklinikum Köln - Klinik I fur Innere Medizin - Klinisches Studienzentrum fur Infektiologie I, Cologne
  - Universitätsklinikum Essen - Klinik fur Dermatologie und Venerologie - HPSTD Ambulanz, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik II, Schwerpunkt Infektiologie, Haus 68, Frankfurt am Main
  - Infektiologikum Frankfurt, Frankfurt am Main
  - ICH Study Center GmbH & Co. KG, Hamburg
  - Universitätsklinikum Hamburg- Eppendorf - Ambulanzzentrum des Universitatsklinikums Eppendorf GmbH - Bereich Infektiologie, Hamburg
- Puerto Rico (4):
  - Instituto de Investigacion Cientifica del Sur, Ponce
  - Hope Clinical Research, San Juan
  - Proyecto ACTU, San Juan
  - Clinical Research Puerto Rico, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Sax PE, Rockstroh JK, Luetkemeyer AF, Yazdanpanah Y, Ward D, Trottier B, Rieger A, Liu H, Acosta R, Collins SE, Brainard DM, Martin H; GS-US-380-4030 Investigators. Switching to Bictegravir, Emtricitabine, and Tenofovir Alafenamide in Virologically Suppressed Adults With Human Immunodeficiency Virus. Clin Infect Dis. 2021 Jul 15;73(2):e485-e493. doi: 10.1093/cid/ciaa988. PMID 32668455
- [Result] Acosta RK, Willkom M, Andreatta K, Liu H, Martin R, Parvangada A, Martin H, Collins S, White KL. Switching to Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) From Dolutegravir (DTG)+F/TAF or DTG+F/Tenofovir Disoproxil Fumarate (TDF) in the Presence of Pre-existing NRTI Resistance. J Acquir Immune Defic Syndr. 2020 Nov 1;85(3):363-371. doi: 10.1097/QAI.0000000000002454. PMID 32701823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 12 June 2017. The last study visit occurred on 10 Feb 2021.
Pre-assignment Details: 633 participants were screened.
Groups:
- B/F/TAF: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed-dose combination (FDC) tablet + dolutegravir (DTG) placebo tablet + emtricitabine/tenofovir alafenamide (F/TAF) placebo tablet administered orally once daily without regard to food for at least 48 weeks.
- DTG + F/TAF: DTG 50 mg tablet + F/TAF (200/25 mg) FDC tablet + B/F/TAF placebo tablet administered orally once daily without regard to food for at least 48 weeks.
- B/F/TAF From B/F/TAF: Participants who received B/F/TAF in double-blind phase and from a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
- B/F/TAF From DTG + F/TAF: Participants who received DTG + F/TAF in double-blind phase and from a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
Period: Double-Blind Treatment Phase
Arm/Group | B/F/TAF | DTG + F/TAF | B/F/TAF From B/F/TAF | B/F/TAF From DTG + F/TAF
Started | 284 | 283 | 0 | 0
Safety Analysis Set | 284 | 281 | 0 | 0
Completed | 263 | 253 | 0 | 0
Not Completed | 21 | 30 | 0 | 0
Not completed — Withdrew Consent | 10 | 16 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 0
Not completed — Investigator's Discretion | 1 | 3 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Non-Compliance with Study Drug | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Randomized but not Treated | 0 | 2 | 0 | 0
Period: Open-label B/F/TAF Extension Phase
Arm/Group | B/F/TAF | DTG + F/TAF | B/F/TAF From B/F/TAF | B/F/TAF From DTG + F/TAF
Started | 0 (Following the end of Double-Blind treatment phase, participants in a country where B/F/TAF FDC was not available were given the option to receive open-label B/F/TAF.) | 0 (Following the end of Double-Blind treatment phase, participants in a country where B/F/TAF FDC was not available were given the option to receive open-label B/F/TAF.) | 125 (138 participants completed the Double-Blind treatment phase, but did not continue in the Open-label B/F/TAF extension phase.) | 116 (137 participants completed the Double-Blind treatment phase, but did not continue in the Open-label B/F/TAF extension phase.)
Completed | 0 | 0 | 121 | 113
Not Completed | 0 | 0 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Withdrew Consent | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- B/F/TAF: B/F/TAF (50/200/25 mg) FDC tablet + DTG placebo tablet + F/TAF placebo tablet administered orally once daily without regard to food for at least 48 weeks.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | DTG + F/TAF | Total
Number analyzed (Participants) | 284 | 281 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.3) | 49 (11.3) | 50 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 245 | 240 | 485
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 3 | 3 | 6
  Race: Black | 68 | 61 | 129
  Race: Native Hawaiian or Pacific Islander | 2 | 1 | 3
  Race: White | 200 | 199 | 399
  Race: Other | 9 | 13 | 22
  Race: Not Permitted | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 61 | 49 | 110
  Ethnicity: Not Hispanic or Latino | 220 | 229 | 449
  Ethnicity: Not Permitted | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 24 | 25 | 49
  Austria | 2 | 1 | 3
  United States | 197 | 202 | 399
  France | 12 | 14 | 26
  Germany | 30 | 26 | 56
  Puerto Rico | 19 | 13 | 32
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 276 | 275 | 551
  ≥ 50 copies/mL | 8 | 6 | 14
CD4 Cell Count [Mean (Standard Deviation); unit: Cells/μL] | 714 (309.1) | 658 (294.7) | 686 (303.1)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 50 Cells/ μL | 0 | 1 | 1
  ≥ 50 to < 200 Cells/μL | 6 | 6 | 12
  ≥ 200 to < 350 Cells/μL | 18 | 34 | 52
  ≥ 350 to < 500 Cells/μL | 53 | 44 | 97
  ≥ 500 Cells/ μL | 207 | 196 | 403

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 284 | 281
percentage of participants | 0.4 | 1.1
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; The null hypothesis was that the B/F/TAF group is at least 4% higher than the DTG + F/TAF group with respect to the percentage of participants with HIV-1 RNA ≥ 50 copies/mL as determined by the US FDA-defined snapshot algorithm at Week 48; the alternative hypothesis was that the B/F/TAF group is less than 4% higher than the DTG + F/TAF group with respect to the percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48; Test type: Non-Inferiority — A sample size of 260 participants per treatment group would provide at least 90% power to detect a non-inferiority margin of 4% in difference in percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 between the two treatment groups. This was based on the assumptions that both treatment groups have 2% of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 (based on Gilead Genvoya and Stribild studies) and that the significance level of the test is at a one-sided 0.025 level; Difference in Percentages = -0.7, 95.001% CI 2-sided [-2.8 to 1.0] — The differences in percentages of participants between treatment groups and their 95.001% confidence intervals (CI) were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Superiority; p = 0.37, Fisher Exact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 284 | 281
percentage of participants | 93.3 | 91.1
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Non-Inferiority — It would be concluded that B/F/TAF is noninferior to DTG+F/TAF if the lower bound of the 2-sided 95.001% CI of the difference between treatment groups (B/F/TAF group -DTG+F/TAF group) in the percentage of participants with HIV-1 RNA < 50 copies/mL is greater than -10%; Difference in Percentages = 2.2, 95.001% CI 2-sided [-2.3 to 6.8] — The differences in percentages of participants between treatment groups and their 95.001% CI were calculated based on an unconditional exact method using 2 inverted 1-sided tests

3. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF | DTG + F/TAF
Number analyzed (Participants) | 262 | 256
cells/µL | 18 (179.1) | 36 (152.6)
Statistical Analysis 1: Comparison: B/F/TAF vs DTG + F/TAF; Test type: Superiority; p = 0.23, ANOVA; P-value, difference in least squares means (LSM), and its 95% CI were from ANOVA model with treatment group as a fixed effect in the model; Difference in LSM = -18, 95% CI 2-sided [-46 to 11]

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date [maximum: 84.9 weeks (Blinded Phase), 179.6 weeks (Open Label Phase) plus 30 days All-Cause Mortality: Randomization/Enrollment up to 187.7 weeks
Description: Adverse Events: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
  All-Cause Mortality: The All Randomized Analysis Set included all participants who were randomized into the study.
Groups:
- Double-Blind Treatment Phase B/F/TAF: B/F/TAF (50/200/25 mg) FDC tablet + DTG placebo tablet + F/TAF placebo tablet administered orally once daily without regard to food for atleast 48 weeks.
- Double-Blind Treatment Phase DTG + F/TAF: DTG 50 mg tablet + F/TAF (200/25 mg) FDC tablet + B/F/TAF placebo tablet administered orally once daily without regard to food for atleast 48 weeks.
- Open-label Extension Phase B/F/TAF From B/F/TAF: Participants who received B/F/TAF in double-blind phase and from a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
- Open-label Extension Phase B/F/TAF From DTG + F/TAF: Participants who received DTG + F/TAF in double-blind phase and from a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
Arm/Group | Double-Blind Treatment Phase B/F/TAF | Double-Blind Treatment Phase DTG + F/TAF | Open-label Extension Phase B/F/TAF From B/F/TAF | Open-label Extension Phase B/F/TAF From DTG + F/TAF
All-Cause Mortality (participants affected / at risk) | 3/284 | 2/283 | 0/125 | 0/117
Serious Adverse Events (participants affected / at risk) | 36/284 | 27/281 | 12/125 | 11/116
Other Adverse Events (participants affected / at risk) | 181/284 | 170/281 | 30/125 | 33/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment Phase B/F/TAF (N=284) | Double-Blind Treatment Phase DTG + F/TAF (N=281) | Open-label Extension Phase B/F/TAF From B/F/TAF (N=125) | Open-label Extension Phase B/F/TAF From DTG + F/TAF (N=116)
Lymphocytic infiltration (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis orbital (Infections and infestations) | 1 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 2
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Yolk sac tumour site unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Vertebral artery dissection (Nervous system disorders) | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 2 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Rebound psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment Phase B/F/TAF (N=284) | Double-Blind Treatment Phase DTG + F/TAF (N=281) | Open-label Extension Phase B/F/TAF From B/F/TAF (N=125) | Open-label Extension Phase B/F/TAF From DTG + F/TAF (N=116)
Diarrhoea (Gastrointestinal disorders) | 26 | 35 | 4 | 7
Fatigue (General disorders) | 22 | 9 | 1 | 7
Bronchitis (Infections and infestations) | 18 | 14 | 4 | 5
Influenza (Infections and infestations) | 19 | 17 | 2 | 1
Nasopharyngitis (Infections and infestations) | 44 | 32 | 3 | 1
Sinusitis (Infections and infestations) | 16 | 11 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 33 | 40 | 9 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 21 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 15 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 15 | 1 | 4
Headache (Nervous system disorders) | 16 | 23 | 1 | 4
Insomnia (Psychiatric disorders) | 19 | 14 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 16 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 15 | 0 | 2
Hypertension (Vascular disorders) | 15 | 11 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03110380/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03110380/SAP_002.pdf